CLINICAL TRIAL: NCT05669781
Title: The Effects of Combined Gum-chewing and Parenteral Metoclopramide on the Duration of Post-operative Ileus After Abdominal Surgery
Brief Title: The Effects of Combined Gum-chewing and Parenteral Metoclopramide on Post-operative Ileus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ikechukwu Bartholomew Ulasi (Other)
Responsible Party: Sponsor-Investigator, Ikechukwu Bartholomew Ulasi, Principal investigator, University College Hospital, Ibadan
Organization: University College Hospital, Ibadan (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: UI/EC/18/0231
Record Dates: First submitted 2022-12-17; First posted 2023-01-03 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Ileus Postoperative
Keywords: Gum-chewing; Metoclopramide; Abdominal; Surgery
MeSH Terms: interventions — Metoclopramide; Chewing Gum

STUDY DESIGN:
Intervention Model Description: Patients were randomized into a gum-metoclopramide (GM) group, a gum-only (G) group, a metoclopramide-only (M) group and a control (C) group. Patients in the GM group chewed gum and received intravenous metoclopramide, each 8 hourly. In the G group, patients chewed only gum while those in the M group received 10mg of intravenous metoclopramide only. To the C group, 10ml of intravenous sterile water for injection was given 8 hourly
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Gum-Metoclopramide (Active Comparator): Intravenous metoclopramide 10mg 8hourly for the first 72hours post-operatively and to chew one a stick of sugar free gum (to be chewed over 15minutes) 8 hourly till either first flatus or feces was passed
  Interventions: Combination Product: Gum and metoclopramide
- Gum-only (Active Comparator): Chew one stick of sugar free gum (to be chewed over 15minutes) 8 hourly till either first flatus or feces was passed
  Interventions: Other: Gum
- Metoclopramide-only (Active Comparator): Intravenous metoclopramide 10mg 8hourly for the first 72hours post-operatively
  Interventions: Drug: Metoclopramide 10mg
- Control (Placebo Comparator): 10ml of sterile water intravenously 8hourly for the first 72hours post-operatively
  Interventions: Other: Control

INTERVENTIONS:
Drug: Metoclopramide 10mg — Intravenous metoclopramide 10mg 8hourly for the first 72hours post-operatively
  Other Names: Philometro, Hubei Tianyao
  Arms: Metoclopramide-only
Combination Product: Gum and metoclopramide — Intravenous metoclopramide 10mg 8hourly for the first 72hours post-operatively and one stick of sugar-free gum (over 15minutes) 8 hourly till either the first flatus or feces was passed
  Arms: Gum-Metoclopramide
Other: Gum — One stick of sugar-free gum (over 15minutes) 8 hourly till either the first flatus or feces was passed
  Arms: Gum-only
Other: Control — 10ml of sterile water intravenously 8hourly for the first 72hours post-operatively
  Arms: Control

SUMMARY:
A delay in the return of bowel function is a common occurrence after abdominal surgeries.1 The goal of this study was to test the effect of the combined use of chewing a gum and administering metoclopramide intravenously on the duration of this natural delay in the return of bowel function after abdominal surgeries. Patients were grouped into four: the first group received both gum and metoclopramide; the second group received only gum; the third group received only metoclopramide, while the fourth group (the control group) received sterile water for injection. The groups were compared for the time taken for bowel function to return and the duration of hospital stay.

DETAILED DESCRIPTION:
This was a prospective randomized controlled trial that recruited all patients requiring elective abdominal surgery, aged 16-65years. Abdominal emergency surgeries and structural or functional inability to chew gum constituted the exclusion criteria. A written informed consent was obtained from all eligible patients.

Considering an effect size of 0.8(Cohen, 1962)2 at a power of 80% with 95% level of confidence and type-1 error of 5%, a total sample size of 105 study participants was obtained, having considered an attrition rate of 5%. Study participants were randomized into 4 groups (a gum-metoclopramide {GM} group, a gum-only {G} group, a metoclopramide-only {M} group and a control {C} group) using blocked sequence randomization.

Data was obtained through a detailed history and physical examination and include demographic variables like age and gender. Medical history of previous abdominal surgeries and any comorbidity like chronic constipation, diabetes mellitus, parkinsonism, renal or cardiac disease were sought and allergy to metoclopramide or gum noted. Body Mass Index (BMI) and relevant investigation results were recorded. Other pre- and intra-operative data recorded included: clinical diagnosis, American Society of Anaesthesiologists (ASA) grade, type of anaesthesia, cadre of surgeon, surgical access (laparoscopic versus open), length of skin incision, intra-operative blood loss, total intra-operative fluid administered, duration of surgery, surgical procedure done and duration of anaesthesia. Recorded post-operatively were time to passage of first flatus, time to passage of first feces, time to initial recording of bowel sounds, time to tolerance of normal diet, day of first ambulation, length of hospital stay, cost of hospital stay and post-operative complications.

Informed consent was obtained from all patients that met the inclusion criteria. All patients for elective surgery were admitted at least a day prior to surgery and kept on nothing by mouth from 12midnight on the eve of surgery. Patients were given intravenous metronidazole and ceftriaxone at the induction of anaesthesia. All the patients had general anaesthesia. Abdominal skin incision was made by the surgeon who was either a senior registrar or consultant in general surgery and to whom the patient's group was undisclosed. Standard procedures (surgical and anesthetic) relevant for each case were carried out. The group assigned to each patient was known only to the research assistants (a house surgeon and the nursing staff) who alone administered the intervention to the appropriate groups. Although what was used for intravenous intervention was undisclosed to the patients in the GM, M and C groups, it was not possible to blind patients who received gum only (G group).

All interventions were commenced from the 1st post-operative day. Patients in the gum-only(G) group were given one stick of sugar free gum (Orbit, Wrigley, US) 3 times 8 hourly daily (in the morning, afternoon and in the evening) till either first flatus or feces was passed with an instruction to chew for 15 minutes(only) without swallowing the chewed gum. The criteria for discontinuing each intervention was not disclosed to the patients. The gum was given to patients at a fixed interval to help monitor compliance. Patients in the metoclopramide-only (M) group received intravenous metoclopramide (Philometro, Hubei Tianyao) 10mg 8hourly for the first 72hours post-operatively. The gum-metoclopramide (GM) group received intravenous metoclopramide and also chewed gum using the protocol earlier described for gum only and metoclopramide only groups. Patients assigned to the control (C) group received 10ml of sterile water intravenously 8hourly for the first 72hours post-operatively.

All patients were asked to notify the nursing staff at first passage of flatus. A blinded doctor visited the patients 8hourly and recorded the time of the first bowel sounds, passage of flatus, and defecation. After giving each intervention, the type and time of intervention was documented in an identifier-free patient's questionnaire. The first time of flatus and defecation was recorded based on the patient's own statements. Prolonged post-operative ileus was defined as ileus lasting more than 5days following laparotomy or greater than 3days following laparoscopic surgery.3 Nasogastric tube was removed on the day of return of bowel function. The total duration of hospital stay, calculated from the first post-operative day to the day of discharge, was recorded.

The association between categorical and numerical peri-operative factors with prolonged post-operative ileus was analyzed using the Chi-square (and Fisher's exact) test and independent t-test (and Mann Whitney-U test) respectively. Comparison of groups in terms of the duration of post-operative ileus and duration of hospital stay was done using analysis of variance (ANOVA). Secondary endpoints compared between the groups included time to first bowel sound, duration of hospital stay and cost of hospital stay. Statistical significance was set at a p-value of <0.05. Version 23 of the Statistical Package for Social Sciences for Windows was used to analyze all data obtained from this study.

ELIGIBILITY:
Inclusion Criteria:

* All patients requiring elective abdominal surgery aged 16-65years

Exclusion Criteria:

* Abdominal emergency surgeries
* Structural or functional inability to chew gum

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Duration of post-operative ileus | From 24 hours after surgery up to the time either flatus or feces is passed, for up to 1week after surgery
  Time to either the passage of flatus or feces, assessed every 8hours from post-operative day 1

SECONDARY OUTCOMES:
Duration of hospital stay | First post-operative day up to the day of discharge, for up to 25days after surgery
  Length of in-hospital care after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ikechukwu B. Ulasi, Principal Investigator — University College Hospital, Ibadan
Locations (1):
- University College Hospital, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pedziwiatr M, Kisialeuski M, Wierdak M, Stanek M, Natkaniec M, Matlok M, Major P, Malczak P, Budzynski A. Early implementation of Enhanced Recovery After Surgery (ERAS(R)) protocol - Compliance improves outcomes: A prospective cohort study. Int J Surg. 2015 Sep;21:75-81. doi: 10.1016/j.ijsu.2015.06.087. Epub 2015 Jul 29. PMID 26231994
- [Background] COHEN J. The statistical power of abnormal-social psychological research: a review. J Abnorm Soc Psychol. 1962 Sep;65:145-53. doi: 10.1037/h0045186. No abstract available. PMID 13880271
- [Background] Delaney C, Kehlet H, Senagore AJ, Bauer AJ, Beart R, Billingham R, et al. Postoperative ileus: profiles, risk factors, and definitions - a framework for optimizing surgical outcomes in patients undergoing major abdominal colorectal surgery. In: Bosker G, editor. Clinical consensus update in general surgery; 2006 May 1; Massachusetts United States. Roswell (GA): Pharmatecture, LLC; 2006. p. 1-26.